CLINICAL TRIAL: NCT00935285
Title: Immune Response in Patients Who Develop Ventilator-Associated Pneumonia (VAP) in Intensive Care Unit (ICU) and the Role of Toll-Like Receptors(TLR2,TLR4,TLR9).
Brief Title: Ventilator-Associated Pneumonia (VAP) in Intensive Care Unit (ICU)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: ZAKYNTHINOS E, INTENSIVE CARE UNIT DEPARTMENT UNIVERSITY HOSPITAL OF LARISA
Other Study IDs: 1692UT
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Ventilator-Associated Pneumonia
Keywords: Ventilator-associated pneumonia (VAP); Intensive care unit (ICU); Toll-like receptors
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Ventilator-associated pneumonia (VAP) is very common in the intensive care unit (ICU), affecting 9 to 40% of ICU patients and mortality rates range from 20 to 50% and may reach more than 70% when the infection is caused by multi-resistant and invasive pathogens. The most common pathogens that cause VAP are the Gram(-) bacteria. Findings indicate that TLRs serves as an important signal in the generation of protective innate responses to bacterial pathogens of the lung and that is required for effective innate immune responses against Gram-negative bacterial pathogens. There is genetic evidence that mutations in TLRs increase the risk of developing nosocomial infections. Understanding the TLR system should offer invaluable opportunity for manipulating host immune responses.

DETAILED DESCRIPTION:
INTRODUCTION

Ventilator-associated pneumonia (VAP) typically refers to nosocomial pneumonia developing 48 hours later from endotracheal intubation and mechanical ventilation.ICU patients who receive mechanical ventilation have 4-fold higher risk of developing pneumonia with a rate of 3% per day after day 7 in the intensive care unit. Several risk factors have been reported to be associated with VAP, including the duration of mechanical ventilation, the presence of chronic pulmonary disease, sepsis, acute respiratory distress syndrome (ARDS), neurological disease and trauma. The immune system defends the host against infection. Protective immunity can be divided into innate and adaptive immunity. The innate immune response evolves as a first defence barrier in the host and mounts an immediate, but nonspecific, immune response to rapidly destroy or limit the invaders. The innate defense mechanisms are the external epithelia, the mucosal surfaces, the cells (NK cells, phagocytes) and the complement system.

Adaptive immunity is a second line defence that includes T (cellular) and B (humoral) cell mediated responses. This is specific, targets only pathogens and not self, and has memory to sustain a long-lasting immunity against reinfection. Although the innate immune system lacks the fine specificity of adaptive immunity it can distinguish self from non self. Innate immune recognition is mediated by a system of germline-encoded receptors named pattern recognition receptors (PRRs) that recognize conserved molecular patterns (pathogen-associated molecular patterns, PAMPs) that are associated with microbial pathogens. These receptors are coupled to signal transduction pathways that control expression of a variety of inducible immune-response genes.

TLRs control both innate and adaptive immune responses. The TLR-induced inflammatory response is dependent on a common signaling pathway that is mediated by the adaptor molecule MyD88. TLR expression is observed in a variety of cells such as macrophages, neutrophils, dendritic cells, epithelial cells derived from gut, lung and derma, B-and T-lymphocytes.TLR4 was the first mammalian TLR identified and is involved in the recognition of lipopolysaccharide (LPS), a major cell wall component of Gram-negative bacteria which can induce sepsis. TLR2 is the most powerful receptor and recognizes a wide variety of PAMPs from bacteria, yeast, fungi, parasites and viruses. TLR9 recognizes unmethylated CpG motifs present in bacterial DNA.

Sepsis syndrome is frequently complicated by the development of nosocomial infections, particularly Gram-negative pneumonia. Findings indicate that TLR9 serves as an important signal in the generation of protective innate responses to bacterial pathogens of the lung and that is required for effective innate immune responses against Gram-negative bacterial pathogens. Unmethylated CpG motifs are prevalent in bacterial but not vertebrate genomic DNA. The recognition of CpG motifs activates host defense mechanisms leading to innate and acquired immune responses. Cells that express TLR-9 are the plasmacytoid dendritic cells (PDCs) and the B cells and as a consequences produce Th1-like proinflammatory cytokines, interferons and chemokines. Activation of TLR-9 induces the production of a) cytokines (IL-12, IL-1, IL-6, IL-8), interferon (IFN)-γ and tumor necrosis factor (TNF-)α which are Th1 proinflammatory cytokines and b) IL-10 and IL-4 which are Th2 proinflammatory cytokines that induce immunosuppression.

Th1 cytokines play a central role in inflammation and activation of macrophages, NK cells and neutrophils. Th2 cytokines inhibit Th1 immune response. This causes a systemic systemic inflammatory response syndrome. Also, toll-like receptors-2 (TLR2) and -4 (TLR4) play a crucial role in chronic obstructive pulmonary disease (COPD). Their activation by LPS of Gram (-) and Gram (+) bacteria leads to activation of neutrophils, NK cells, T-, B- cells and inflammatory cytokines. In chronic disease, dysregulated inflammation maintains these systems in a state of constant activation, potentially resulting in tissue damage and progressive disease. Understanding the TLR system should offer invaluable opportunity for manipulating host immune responses.

AIMS

1. To investigate and elucidate the role of CD4+ και CD8+ Τ lymphocytes in pathogenesis of VAP. Also, the level of cytokines IL-4 and IFN-γ the time when the patients in ICU develop VAP and the changes to the subpopulations of Τ lymphocytes.
2. To evaluate apoptosis of macrophages and their capacity to phagocyte in VAP patients.
3. To study the expression and possible polymorphisms of TLR-2, TLR-4 and TLR-9 genes.

Understanding of immune response to VAP will allow the preparation of immunotherapy protocols so as to regulate immunological response.

METHODS

MATERIALS AND METHODS

Bronchoalveolar lavage processing

At the first day, in each patient samples of blood, bronchoalveolar lavage (BAL) and tracheobronchial aspirate (TBA) will be taken. Bronchoscopy is a technique of visualizing the inside of the airways for diagnostic and therapeutic purposes. A bronchoscope is inserted into the airways, usually through the nose or mouth, or occasionally through a tracheostomy. This allows the practitioner to examine the patient's airways for abnormalities such as foreign bodies, bleeding, tumors, or inflammation. Specimens may be taken from inside the lungs: biopsies, fluid (bronchoalveolar lavage), or endobronchial brushing. BAL is typically performed to diagnose lung disease. In particular, BAL is commonly used to diagnose infections in people with immune system problems, pneumonia in people on ventilators and some types of lung cancer. BAL is often used in immunological research as a means of sampling cells or pathogen levels in the lung (T-cell populations). Specimens may be taken again in 48 hours from the diagnosis of VAP. BAL will be placed in 10%FBS-RPMIc and centrifuges at 400g, 5 min, and then will be added RPMI-1640 and 10% FBS. The number and the type of the cells will be defined by Μay-Grunwald-Giemsa staining, and the subpopulations with flow cytometry.

PBMC isolation

Human lymphocytes can be isolated most readily from peripheral blood by density centrifugation with the carbohydrate polymer Ficoll (Ficoll Histopaque, Sigma, Cat 1077-1). This yields a population of mononuclear cells at the interface that has been depleted of red blood cells and most polymorphonuclear leukocytes or granulocytes. The resulting population, called peripheral blood mononuclear cells, consists mainly of lymphocytes and monocytes. Diluted anticoagulated blood is layered over Ficoll and centrifuges at 400g, 30min at 20ºC (slow acceleration, no brake). Red blood cells, polymorphonuclear leukocytes or granulocytes have higher density from Ficoll and are to the bottom of the tube. But mononuclear cells consisting of lymphocytes together with some monocytes band over it and can be recovered at the interface. Cells are washed using 1xPBS with 1mM EDTA 3 times to remove Ficoll and platelets.

Antibody labeling

Anti-CD3-FITC (fluorescein isothiocyanate), anti-CD8-PE (phycoerythrin), anti-CD4-PE, anti-IFN-γ and anti-IL-4, anti-CD4, anti-CD8 and controls IgG-FITC and -PE will be used for labeling cells. Fluorescein isothiocyanate (FITC) a reactive derivative of fluorescein, has been one of the most common fluorophores chemically attached to other, non-fluorescent molecules to create new fluorescent molecules for a variety of applications. DAKO system will be used. For staining, immunochemistry will be used after plating the cells on Superfrost Plus slides by cytocentrifugation with the kit of DAKO according to instructions of the manufacturer.

Immunohistochemistry

Lymphocytes will be stimulated in 24-well plates in RPMI-1640 at 10% fetal calf serum in the presence of phorbol 12-myristate 13 acetate, 25 ng/mL; ionomycin; 1 µmol; and Brefeldin A, 10 µg/mL (Sigma-Aldrich; St, Louis, MO). Cytospins will be made using cytocentrifugation of 150 µL of the stimulated suspension and store at - 80°C. Approximately 175,000 cells will be cytospun on each slide of which are sufficient lymphocytes to stain. The double immunocytochemical method for the determination and measurement of CD8+IFN-+, CD8+IFN-+ (or CD4+IFN-+, CD4+IFN-+) will be performed in two steps. At step one, use the primary anti-CD8 (or anti-CD4, respectively) mouse anti-human monoclonal antibody with secondary rabbit anti-mouse IgG-FITC antibody. At step two, after permeabilization, a primary anti-IFN- or IL-4 mouse anti-human monoclonal antibody (Caltag; Burlingame, CA) with secondary rabbit anti-mouse IgG-PE. A permeabilization kit of will be used according to the instructions of the manufacturer (Dako). For the estimation of each ratio, 500 T cells we count > 10 cytospins stained if necessary because this number is sufficient to obtain a mean value per subject that remain constant after further increasing the number of cells counted.

Flow Cytometric Analysis

The samples prepared as described above were analyzed on a fluorescence activated cytometer (EPICS ELITE; Coultronics; Louton, UK). The lymphocytes were tightly gated by volume and complexity on a forward (0o) and side light scattering (90o) mode. Phycocyanate-conjugated anti-human CD45 monoclonal antibodies (DAKO; Ely, UK) will be used as pan-leukocyte stain to exclude non leukocyte events by logical gating. The percentage of one-color, two-color, and three-color positive cells will be measured and the mean channel value as well as the relative fluorescence intensity (RFI) corresponding to the antigen density wii be estimated. QC-Combo Kit (FCSC; San Jun, Puerto Rico) will be used for the quantification of antibody binding.

Statistical Analysis

Normality of the numerical parameters will be tested using the Kolmogorov-Smirnov test. Wilcoxon signed-rank test for nonparametric outcomes and paired t test for parametric outcomes will be used for comparison of data at two different time points (at stable condition and at exacerbation). Statistical software (SPSS version 11.0; SPSS; Chicago, IL) will be used for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Presence in intensive care unit receive mechanical ventilation <48h have no history of ΑRDS or other respiratory disease

Exclusion Criteria:

* Length of stay <24 hours

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include ICU patients who receive mechanical ventilation <48h and have no history of ΑRDS or other respiratory disease.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Sarafi RN MSc, ICU, Principal Investigator — University Hospital Larisa
Locations (1):
- Zakynthinos, Larissa, Mezourlo, Greece